CLINICAL TRIAL: NCT03612765
Title: The Effectiveness of the Push-Pull-Hold Program on Improving Self-Care in Patients With Heart Failure: A Randomised Controlled Trial
Brief Title: The Effectiveness of the Push-Pull-Hold Program on Improving Self-Care in Patients With Heart Failure
Acronym: PPHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: National Heart Centre Singapore (Other)
Responsible Party: Principal Investigator, Jocelyn Chew, Principal Investigator, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 201804-00157; NTEC-2018-0265 (Other: The Joint CUHK-NTEC CREC)
Record Dates: First submitted 2018-07-19; First posted 2018-08-02 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Heart Failure
Keywords: heart failure; self-care; behavio*; intervention; randomized controlled trial
MeSH Terms: conditions — Heart Failure | interventions — 5-phenylpent-4-enyl-1-hydroperoxide

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group will receive face-to-face intervention sessions that include interviews, discussions and didactic teaching.
  Interventions: Behavioral: Push-Pull-Hold Program
- Control group (No Intervention): Participants in the control group will receive usual care that normally includes three monthly outpatient doctor consultations and when necessary, heart failure nurse referral.

INTERVENTIONS:
Behavioral: Push-Pull-Hold Program — Developed based on concepts of motivational interviewing, temporal framing, empowerment. It is tailored to Singaporean patients and includes contextual self-care information and tips.
  Other Names: PPHP
  Arms: Intervention group

SUMMARY:
This study is a randomized controlled trial that tests the effectiveness of a novel intervention called the Push-Pull-Hold program on improving self-care in patients with heart failure. This intervention was developed based on our previous quantitative and qualitative findings and existing psychological concepts. Results would inform current understanding of the intention-behavior link in self-care and inform future policy and intervention development to improve patient and caregiver outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with chronic heart failure for at least 1 month
* More than 21 years old
* Able to read and understand English or Chinese

Exclusion Criteria:

* Dependent on caregivers
* Awaiting implantable devices or surgery
* Pregnant

Ages: 21 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in Self-Care of Heart Failure Index (SCHFI) maintenance subscale | weeks 1, 12 and 24
  SCHFI maintenance subscale is a 10-item, self-administered instrument that measures self-care maintenance behaviours such as medication adherence. Each item of the instrument is rated on a 4-point Likert scale and each subscale score is rescaled to range from 0 to 100 where a score of more than or equal to 70 represents adequate self-care.

SECONDARY OUTCOMES:
Changes in the Consideration of Future Consequences Scale (CFCS) | weeks 1, 12 and 24
  CFCS is a 14-items self-administered instrument that measures the degree to which one considers about and is influenced by the potential consequences of their present behaviours. Each item is measured using a 7-point Likert scale where 1 represents extremely uncharacteristic and 7 represents extremely characteristic of the participant. The average scores of the items will be calculated, where a higher score indicates a higher consideration of future consequences.
Changes in intention to change behaviours | weeks 1, 12 and 24
  Intention will be measured using a self-developed 3-item, self-administered instrument. Responses will be measured on a 7-point Likert scale where a higher score indicates a higher intention to change behaviours.
Changes in the Self-Report Habit Index (SRHI) | weeks 1, 12 and 24
  SRHI is a 12-items, self-administered instrument that measures automaticity; behaviour frequency; and self-identity on a 7-point Likert scale. Scores will be averaged and a higher score indicates higher habit strength.
Changes in Mindfulness Attention Awareness Scale (MAAS) | weeks 1, 12 and 24
  MAAS is a 15-items, self-administered instrument measured on a 6-point Likert scale. A mean score will be computed and a higher score indicates higher level of mindfulness.
Minnesota Living with Heart Failure Questionnaire (MLHFQ) | weeks 1, 12 and 24
  MLHFQ is a 21-items, self-administered instrument measured on a 6-point Likert scale and includes components of physical, emotional, social and mental dimensions of quality of life. Scores will be summed up and ahigher score indicates poorer quality of life.

OTHER OUTCOMES:
Changes in readmission | Weeks 1 and 24
  Measures the changes in readmission incidences.
Changes in emergency department visits | Weeks 1 and 24
  Measures the changes in the incidence of emergency department visits.
Mortality | Week 24
  Incidence of mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Jocelyn H.S. Chew, BSc(Nursing), Principal Investigator — The Nethersole School of Nursing
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore